CLINICAL TRIAL: NCT01366599
Title: Cardiovascular Events in Cancer Patients Receiving Highly Emetogenic or Moderately Emetogenic Chemotherapy
Brief Title: CV Events in Emetogenic Chemotherapy
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115777; WEUKSTV4114 (Other: GSK)
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Vomiting; Cardiovascular Event; Arterial Thromboembolic Event
Keywords: highly emetogenic chemotherapy; HEC; moderately emetogenic chemotherapy; MEC
MeSH Terms: conditions — Vomiting | interventions — NDC80 protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients enrolled in IHCIS in 2006: Patients enrolled in IHCIS in 2006
  Interventions: Drug: HEC or MEC

INTERVENTIONS:
Drug: HEC or MEC — Any HEC or MEC, including aprepitant

SUMMARY:
Describe cardiovascular events in a cancer population receiving highly emetogenic chemotherapy (HEC) or moderately emetogenic chemotherapy (MEC).

DETAILED DESCRIPTION:
Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymised and used to develop a patient cohort. All diagnoses and treatment are recorded in the course of routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in IHCIS in 2006
* At least one HEC or MEC claim in 2006

Exclusion Criteria:

* HEC or MEC claim three months before first HEC/MEC claim - "wash-in" period (i.e. must be enrolled for three months prior to first HEC/MEC claim. For patients whose first HEC/MEC event is between January 1,2006 and March 31, 2006, enrollment criteria for inclusion in the study may extend as far back as October 1, 2005)
* HEC or MEC claims prior to 45 days after last HEC or MEC claim - "wash-out" period. (For patients whose last claim in 2006 was seen after December 1, 2006 enrollment into 2007 to look for further treatment and the 45 day "wash-out" period will be required.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IHCIS, 2005-2007. The Impact National Managed Care Benchmark Database™ (formally known as Integrated Healthcare Information Services - IHCIS - prior to its purchase by Ingenix, Inc and referred to as IHCIS within GSK) is a comprehensive, de-identified U.S. healthcare claims database that is representative of the non-elderly, insurance-carrying population in the U.S. The database contains inpatient/outpatient and pharmacy claims, lab results and enrollment information on over 82 million lives from 1997 to 2007. Over 75 percent of all patients in the database have both medical and pharmacy benefits and, on average, 23.4 months of enrollment/claims information; the annual attrition rate is roughly 15-25 percent. The data are collected from over 45 different healthcare plans serving members across nine census regions. The database is HIPAA compliant and features encrypted member and provider IDs.
Sampling Method: Non-Probability Sample
Enrollment: 12058 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Calculate the frequency and percent of patients with selected cardiovascular and arterial thromboembolic events in the analysis period, stratifying by any use of aprepitant (Emend) during the analysis period. | First day of first HEC/MEC cycle to 30 days past first day of last cycle